CLINICAL TRIAL: NCT03628768
Title: Risk Factors for Falls and Neurocognitive Disorders in the Older Canadian Population: A Population-based Cross-sectional Study
Brief Title: Risk Factors for Falls and Neurocognitive Disorders CLSA
Status: Active, not recruiting | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, Professor of Geriatrics, Jewish General Hospital
Other Study IDs: 2019-1453
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Neurocognitive Disorders; Geriatrics
MeSH Terms: conditions — Neurocognitive Disorders | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Healthy / Non fallers: Older cognitively healthy individuals Non fallers
  Interventions: Other: Data collection
- Healthy / Fallers without injuries: Older cognitively healthy individuals Fallers without injuries
  Interventions: Other: Data collection
- Healthy / Fallers with injuries: Older cognitively healthy individuals Fallers with injuries
  Interventions: Other: Data collection
- MCI / Non fallers: Older individuals with MCI and mild dementia Non fallers
  Interventions: Other: Data collection
- MCI / Fallers without injury: Older individuals with MCI and mild dementia Fallers without injuries
  Interventions: Other: Data collection
- MCI / Fallers with injury: Older individuals with MCI and mild dementia Fallers with injuries
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — telephone interview questionnaire, in-home face-to-face interview, and data from the Collection Site

SUMMARY:
The study evaluates the association between the neurocognitive decline and falls.

DETAILED DESCRIPTION:
Falls in older adults are a major Canadian public health concern because: 1) They have a high prevalence and incidence (e.g., up to 30% each year in Canada, regardless the cognitive status of fallers), 2) They negatively impact an individual's health condition (e.g., hip fracture) and quality of life (e.g., social withdraw), and 3) They impose a high financial burden on the Canadian health care system (e.g., $2 billion per year). Major neurocognitive disorders are strongly associated with falls and their adverse outcomes. There is a greater risk for falls and fall-related injuries in cognitively impaired individuals, more than doubled compared to cognitively healthy individuals (CHI). The nature of the interactions between neurocognitive disorders and the other risk factors for falls and fall-related injuries are still a matter of debate. For instance, the presence of specific patterns (i.e., types and combinations) of risk factors for falls and fall-related injuries associated with neurocognitive disorders at their onset (i.e., mild cognitive impairment [MCI] and mild dementia) compared to CHI is questioned. Recently, the investigators howed that the identification of risk factors for falls is influenced by the method of data analysis used. The investigators demonstrated that emerging modeling techniques such as artificial neural networks (ANNs) improve the performance criteria of fall prediction compared to classical linear models. Other methods such as Factor Mixture Models (FMMs) may also be helpful in identification of patterns of risk factors for falls and fall-related injuries associated with neurocognitive disorders. Using baseline data from the Canadian Longitudinal Study on Aging (CLSA), the investigator will examine the patterns (i.e., types and combinations) of risk factors for falls and fall-related injuries associated with neurocognitive disorders at their onset by 1) Examining the epidemiology of falls and fall-related injuries, and 2) Modeling and comparing the associations of risk for falls and fall-related injuries between cognitively healthy and impaired (i.e., MCI and mild dementia) older adults participating in the CLSA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 and
* Participants of the Comprehensive CLSA (i.e., individuals who participated in a 90-minute in-home face-to-face interview, and a visit to one of 11 Data Collection Sites across Canada where they took part in a range of physical assessments).

Exclusion Criteria:

* A fall resulting from acute medical events and/or external force,
* Moderate to severe dementia (estimated from performance on cognitive tests and scores of the Activity of Daily Living (ADL) and Instrumental Activity Daily Living (IADL) scales. Abnormal scores will be defined as 2 Standard Deviations (SDs) or more below the normal score of all cognitive tests associated with scores of ADL (/6) <3 and a score of IADL (/8) <4)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Individuals eligible for this study will be the participants of the CLSA
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Fall-related injury | around 12 months
  Fall-related injury is an event which results in a person coming to rest accidentally on the ground or floor. If participants report having had at least one injury during the past 12 month, they will be asked to answer additional questions that are related to the consequence of fall injury.

SECONDARY OUTCOMES:
Medication | around 12 months
  By using a questionnaire all participants will be ask to report the number of medications that they took the preceding month.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No